CLINICAL TRIAL: NCT00222846
Title: Enhancing Adherence in Type 2 Diabetics
Brief Title: Enhancing Adherence in Type 2 Diabetes: The ENHANCE Study
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Mary Ann Sevick, ScD, RN, School of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NIH-R01-NR008792
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Nephropathy
Keywords: Clinical trial; Behavioral research; Patient compliance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Patient Compliance | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Attention control
  Interventions: Behavioral: Attention control
- B (Experimental): Intervention
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Attention control — Participants attend 3 educational seminars, receive a lay diabetes journal, pedometer, and glucose monitoring supplies.
  Arms: A
Behavioral: Intervention — Behavioral intervention of diabetes self-management paired with PDA-based monitoring of dietary intake and physical activity. Participants also receive a pedometer and glucose self-monitoring supplies.
  Arms: B

SUMMARY:
This randomized study will test a behavioral intervention, based on social cognitive theory (SCT), to improve regimen adherence in three different groups of people with type 2 diabetes; (1) those with well controlled blood glucoses and no concurrent chronic renal insufficiency, (2) those with less well-controlled glucoses and no chronic renal insufficiency, and (3) those with chronic renal insufficiency regardless of glucose control. The primary aims of this study are to: (1)determine whether the intervention improves behavioral adherence to the diabetes self-management regimen including dietary adherence, physical activity, and capillary glucose self-monitoring; (2)determine whether the intervention improves clinical outcomes; (3) explore the extent to which self-efficacy is a mediator of adherence,(4) explore the extent to which the effectiveness of the intervention varies with respect to glycemic control and nephrovascular complications at baseline, and (5)explore the impact of a variety of covariates on the effectiveness of the intervention.

Hypothesis #1 is that intervention group participants will perform better than attention control group participants on various measures of adherence to the diabetes management regimen. Primary adherence variables will be dietary intake, and physical activity. Hypothesis #2 is that intervention group participants will have lower HbA1c levels than attention control group participants.

DETAILED DESCRIPTION:
This randomized study, the ENHANCE Study (Enhancing Adherence to Diabetes Self-Management) will test a behavioral intervention, based on social cognitive theory (SCT), to improve regimen adherence in three different groups of people with type 2 diabetes; (1) HbA1c < 8% and no concurrent chronic renal insufficiency, (2) HbA1c>8% and no chronic renal insufficiency, and (3) those with evidence of chronic renal insufficiency regardless of glucose control.

The primary aims of this study are to:

1. . Determine whether the intervention improves behavioral adherence to the diabetes self-management regimen including: 1.a. dietary adherence, as measured by self-report using dietary recalls and the Nutrient Data System, 1.b. physical activity as measured by the CHAMPS Physical Activity Questionnaire as well as pedometer readings, and 1.c. adherence to capillary glucose self-monitoring as assessed by the FreeStyle monitor.
2. . Determine whether the intervention improves clinical outcome measures including: 2.a. glycosylated hemoglobin levels (HbA1c), 2.b. weight loss, 2.c. anthropometrics.
3. . Explore the extent to which self-efficacy is a mediator of adherence.
4. . Explore the extent to which the effectiveness of the intervention varies with respect to glycemic control and nephrovascular complications at baseline.
5. . Explore the impact of a variety of covariates (medications, depression, social support, severity of disease, and general health and sociodemographic characteristics, clinic from which they were recruited, health literacy, and trust in research) on the effectiveness of the intervention.

Hypothesis #1 is that intervention group participants will perform better than attention control group participants on various measures of adherence to the diabetes management regimen. Primary behavioral adherence variables will be dietary intake, and physical activity. Hypothesis #2 is that intervention group participants will have lower HbA1c levels than attention control group participants.

The 6-month intervention includes group classes, held weekly during months 1&2, biweekly during months 3&4, and monthly during month 5&6. Classes focus on building a sense of mastery over the diabetes regimen and features the use of PDA-base dietary self-monitoring. Intervention group participants are compared to an attention care group, that receives monthly contacts. Measurements are made at baseline, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria: Study subjects will include those with: type 2 diabetes mellitus defined according to the 1997 ADA criteria and age of 18 years or greater. We will sample from three different patient populations: (1) 96 individuals who have HbA1c < 8%, and no evidence of chronic renal insufficiency (a serum creatinine <1.3mg/dl for women and <1.5mg/dl for men). (2) 96 individuals with HbA1c > 8%, and no evidence of chronic renal insufficiency, and (3) 96 individuals with evidence of chronic renal insufficiency (a serum creatinine >1.3mg/dl for women and >1.5mg/dl for men, but who have not yet progressed to dialysis), regardless of HbA1c level.

-

Exclusion Criteria: Exclusion criteria were selected to enhance safety and ability to complete the study protocol. They include: (1) history of hypoglycemic coma/seizure within the last 12 months, (2) hypoglycemia requiring 3rd party assistance within the last 3 months, (3) history consistent with type 1 diabetes, (4) unwillingness to do capillary blood testing using the FreeStyle monitor, (5) unwillingness or inability to participate in scheduled group classes or individual counseling sessions, (7) subjects currently on renal dialysis, (8) any factors likely to preclude adherence to the study protocol including dementia, alcohol or substance abuse, plan to move within the next 8 months, lack of support from the subject's primary health care provider (i.e. PCP is aware of significant risks such as extreme variation in blood glucoses and/or comorbidities that would make participation in the study unsafe), failure to obtain informed consent from the participant, current participation in another clinical trial, and (9) subjects who are not available by telephone during the hours of 8am to 6pm.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2004-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Physical activity CHAMPS | Baseline, 3 and 6 months
Glycemic control - HbA1c | Baseline, 3 and 6 months
Dietary adherence | Baseline, 3 and 6 months

SECONDARY OUTCOMES:
Adherence to capillary glucose checks - glucometer uploads | Baseline, 3 and 6 months
Weight loss | Baseline, 3 and 6 months
BMI | Baseline, 3 and 6 months
Waist circumference | Baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Sevick, ScD, RN, Principal Investigator — University of PIttsburgh & Veterans Health Administration
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Sevick MA, Korytkowski M, Stone RA, Piraino B, Ren D, Sereika S, Wang Y, Steenkiste A, Burke LE. Biophysiologic outcomes of the Enhancing Adherence in Type 2 Diabetes (ENHANCE) trial. J Acad Nutr Diet. 2012 Aug;112(8):1147-57. doi: 10.1016/j.jand.2012.05.008. PMID 22818724